CLINICAL TRIAL: NCT06103305
Title: Risk Stratifications for Patients Come With Palpitations in Assiut and Suez Canal University Hospitals
Brief Title: Risk Stratifications for Patients With Palpitations
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Zakaria Farah Tawdros, Resident physician, Assiut University
Other Study IDs: palpitations
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmias, Cardiac
Keywords: palpitations
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of the study is to early diagnose and early proper mangment of those patients who have palpitations specially of cardiac origin

DETAILED DESCRIPTION:
Palpitation : are one of the most common presentations to general practice, and while they are usually benign, they may also have life-threatening significance. Palpitations have been estimated to account for 16% of general practice presentations and are the second most common presentation to cardiologists after chest pain.

ELIGIBILITY:
Inclusion Criteria:

The present study will be conducted on patients with Palpitations "without intently selected certain gender" and had 18 years old or more

Exclusion Criteria:

patients refusing study will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from 18 years old to 80 years old come to emergency department with palpitations
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality during 30 days follow up

SECONDARY OUTCOMES:
Hospital admission | 0 days
  Admission to hospital from the Emergency Department
ICU admission | 0 days
  Admission to the Intensive Care Unit or High Dependency Unit from the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa Ahmed Herdan, professor, Study Director — Assiut University; Monira Taha ismail, professor, Study Director — Suez Canal University; Hany El moraba, professor, Study Director — Assiut University

REFERENCES:
- [Background] Giada F, Inama G, Bertaglia M, Pedrinazzi C, Gulizia M, Ricci R, Raviele A; Associazione Italiana di Aritmologia e Cardiostimolazione. [Management of patients with palpitations. Consensus document of the AIAC (Italian Association of Arrhythmiology and Cardiostimulation]. G Ital Cardiol (Rome). 2010 Apr;11(4):329-40. No abstract available. Italian. PMID 20677582
- [Background] Probst MA, Mower WR, Kanzaria HK, Hoffman JR, Buch EF, Sun BC. Analysis of emergency department visits for palpitations (from the National Hospital Ambulatory Medical Care Survey). Am J Cardiol. 2014 May 15;113(10):1685-90. doi: 10.1016/j.amjcard.2014.02.020. Epub 2014 Mar 1. PMID 24698469
- [Background] Weber BE, Kapoor WN. Evaluation and outcomes of patients with palpitations. Am J Med. 1996 Feb;100(2):138-48. doi: 10.1016/s0002-9343(97)89451-x. PMID 8629647
- [Background] Lessmeier TJ, Gamperling D, Johnson-Liddon V, Fromm BS, Steinman RT, Meissner MD, Lehmann MH. Unrecognized paroxysmal supraventricular tachycardia. Potential for misdiagnosis as panic disorder. Arch Intern Med. 1997 Mar 10;157(5):537-43. PMID 9066458
- [Background] Porter MJ, Morton JB, Denman R, Lin AC, Tierney S, Santucci PA, Cai JJ, Madsen N, Wilber DJ. Influence of age and gender on the mechanism of supraventricular tachycardia. Heart Rhythm. 2004 Oct;1(4):393-6. doi: 10.1016/j.hrthm.2004.05.007. PMID 15851189
- [Background] Gale CP, Camm AJ. Assessment of palpitations. BMJ. 2016 Jan 6;352:h5649. doi: 10.1136/bmj.h5649. No abstract available. PMID 26739319
- [Background] Dixit S, Stein PK, Dewland TA, Dukes JW, Vittinghoff E, Heckbert SR, Marcus GM. Consumption of Caffeinated Products and Cardiac Ectopy. J Am Heart Assoc. 2016 Jan 26;5(1):e002503. doi: 10.1161/JAHA.115.002503. PMID 26813889
- [Background] Ng GA. Treating patients with ventricular ectopic beats. Heart. 2006 Nov;92(11):1707-12. doi: 10.1136/hrt.2005.067843. No abstract available. PMID 17041126
- [Background] Reddy RK, Pooni R, Zaharieva DP, Senf B, El Youssef J, Dassau E, Doyle Iii FJ, Clements MA, Rickels MR, Patton SR, Castle JR, Riddell MC, Jacobs PG. Accuracy of Wrist-Worn Activity Monitors During Common Daily Physical Activities and Types of Structured Exercise: Evaluation Study. JMIR Mhealth Uhealth. 2018 Dec 10;6(12):e10338. doi: 10.2196/10338. PMID 30530451
- [Background] Raviele A, Giada F, Bergfeldt L, Blanc JJ, Blomstrom-Lundqvist C, Mont L, Morgan JM, Raatikainen MJ, Steinbeck G, Viskin S, Kirchhof P, Braunschweig F, Borggrefe M, Hocini M, Della Bella P, Shah DC; European Heart Rhythm Association. Management of patients with palpitations: a position paper from the European Heart Rhythm Association. Europace. 2011 Jul;13(7):920-34. doi: 10.1093/europace/eur130. No abstract available. PMID 21697315
- [Background] Thavendiranathan P, Bagai A, Khoo C, Dorian P, Choudhry NK. Does this patient with palpitations have a cardiac arrhythmia? JAMA. 2009 Nov 18;302(19):2135-43. doi: 10.1001/jama.2009.1673. PMID 19920238
- [Background] Voskoboinik A, Prabhu S, Ling LH, Kalman JM, Kistler PM. Alcohol and Atrial Fibrillation: A Sobering Review. J Am Coll Cardiol. 2016 Dec 13;68(23):2567-2576. doi: 10.1016/j.jacc.2016.08.074. PMID 27931615
- [Background] Flannery MD, Kalman JM, Sanders P, La Gerche A. State of the Art Review: Atrial Fibrillation in Athletes. Heart Lung Circ. 2017 Sep;26(9):983-989. doi: 10.1016/j.hlc.2017.05.132. Epub 2017 Jun 3. PMID 28606607
- [Background] Flaker GC, Belew K, Beckman K, Vidaillet H, Kron J, Safford R, Mickel M, Barrell P; AFFIRM Investigators. Asymptomatic atrial fibrillation: demographic features and prognostic information from the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):657-63. doi: 10.1016/j.ahj.2004.06.032. PMID 15990749
- [Background] Blomstrom-Lundqvist C, Scheinman MM, Aliot EM, Alpert JS, Calkins H, Camm AJ, Campbell WB, Haines DE, Kuck KH, Lerman BB, Miller DD, Shaeffer CW Jr, Stevenson WG, Tomaselli GF, Antman EM, Smith SC Jr, Alpert JS, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Hiratzka LF, Hunt SA, Jacobs AK, Russell RO Jr, Priori SG, Blanc JJ, Budaj A, Burgos EF, Cowie M, Deckers JW, Garcia MA, Klein WW, Lekakis J, Lindahl B, Mazzotta G, Morais JC, Oto A, Smiseth O, Trappe HJ; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines. Writing Committee to Develop Guidelines for the Management of Patients With Supraventricular Arrhythmias. ACC/AHA/ESC guidelines for the management of patients with supraventricular arrhythmias--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Supraventricular Arrhythmias). Circulation. 2003 Oct 14;108(15):1871-909. doi: 10.1161/01.CIR.0000091380.04100.84. No abstract available. PMID 14557344